CLINICAL TRIAL: NCT02071160
Title: Melatonin for Neuroprotection Following Perinatal Asphyxia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Mahdy, Assistant Professor of Pediatrics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01012012
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Perinatal Asphyxia
Keywords: HIE; hypothermia; encephalopathy; anti oxidants; MRI
MeSH Terms: conditions — Hypothermia; Brain Diseases | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Control (No Intervention): A group of healthy control without any history suggestive of perinatal asphyxia or other diseases, are enrolled to compare different laboratory measurements
- Hypothermia Group (No Intervention): HIE infants who will not receive melatonin and only receive routine cooling protocol.
- Melatonin/ hypothermia group (Experimental): HIE infants who will receive melatonin in addition to the routine cooling protocol
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin is administered to the melatonin/hypothermia group (n=15) in a dose of 10 mg/kg daily for a total of 5 doses starting immediately at enrollment. Melatonin tablets (1 or 3 mg/tablet) (Puritan's Pride,Oakdale, NY, USA) are crushed, then dissolved in 5-10 ml of distilled water , then administered via an orogastric tube.
  Arms: Melatonin/ hypothermia group

SUMMARY:
The aim of this study is to examine the effect of combining melatonin to whole body cooling on the brain injury and outcome of neonates following perinatal asphyxia.

DETAILED DESCRIPTION:
This is a prospective study on 30 neonates with moderate to moderately to severe hypoxic ischemic encephalopathy (HIE) . HIE infants are randomized into two groups: Whole body cooling group (N = 15; receive 72 hours of whole body hypothermia) and melatonin/ hypothermia group (N = 15; receive hypothermia and 5 daily enteral doses of melatonin 10 mg/kg). Serum melatonin, plasma superoxide dismutase (SOD),and serum nitric oxide (NO) are measured at enrollment and after 2 weeks for the two HIE groups. The HIE groups underwent electroencephalography at enrollment and at 2 to 3 weeks. Brain MRI was performed after 2 weeks of life. Neurologic evaluations and Denver Developmental Screening Test II assessments were performed at 6 months. A group of healthy newborns will be used as a control for baseline labs.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants at term gestation (38-42 weeks)
* Apgar scores ≤ 3 at 5 minutes and/or delayed first breath (>5 minutes after birth)
* Profound metabolic or mixed acidosis with serum bicarbonate levels of <12 mmol/L in initial blood gas analyses
* Evidence of moderate or moderate to severe encephalopathy, such as lethargy, seizures, abnormal reflexes, or hypotonia, in the immediate neonatal period

Exclusion Criteria:

* Twin gestation
* Maternal neuro-endocrinal disturbances including diabetes mellitus
* Chorioamnionitis or congenital infections
* Low birth weight less than 2.5 kg
* Congenital malformations of the central nervous system or gastrointestinal anomalies
* Chromosomal abnormalities
* After 6 hours of birth.
* Patients in extremis such as: (1) hypoxemia requiring supplemental oxygen 100% FiO2, (2) life threatening coagulopathy, or (3) deep coma.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Serum melatonin concentration (pg/ ml) | 5 days
Plasma superoxide dismutase (SOD) activity (U/ml) | 5 days
Serum nitric oxide (NO) concentrations (µmol/L) | 5 days

SECONDARY OUTCOMES:
Incidence of EEG abnormalities | 2 weeks
Incidence of MRI abnormalities | 2 weeks
Incidence of abnormal neurological examination | 6 months
Incidence of abnormal Denver Developmental Screening Test II | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heba Mahdy, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta University Children's Hospital, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Gitto E, Reiter RJ, Cordaro SP, La Rosa M, Chiurazzi P, Trimarchi G, Gitto P, Calabro MP, Barberi I. Oxidative and inflammatory parameters in respiratory distress syndrome of preterm newborns: beneficial effects of melatonin. Am J Perinatol. 2004 May;21(4):209-16. doi: 10.1055/s-2004-828610. PMID 15168319
- [Background] Gitto E, Romeo C, Reiter RJ, Impellizzeri P, Pesce S, Basile M, Antonuccio P, Trimarchi G, Gentile C, Barberi I, Zuccarello B. Melatonin reduces oxidative stress in surgical neonates. J Pediatr Surg. 2004 Feb;39(2):184-9; discussion 184-9. doi: 10.1016/j.jpedsurg.2003.10.003. PMID 14966737
- [Background] Chen YC, Tain YL, Sheen JM, Huang LT. Melatonin utility in neonates and children. J Formos Med Assoc. 2012 Feb;111(2):57-66. doi: 10.1016/j.jfma.2011.11.024. Epub 2012 Feb 15. PMID 22370283